CLINICAL TRIAL: NCT04870827
Title: The Effect of Chronic Inflammation on Myocardial Perfusion and Function
Brief Title: Effect of Chronic Inflammation on Myocardial Perfusion and Function
Status: Terminated | Type: Observational
Why Stopped: PI left NIH, study won't meet it's study aims, so closing study.
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 10000136; 000136-H
Record Dates: First submitted 2021-05-01; First posted 2021-05-04 (Actual); Last update posted 2023-04-06 (Actual); Status verified 2023-03

CONDITIONS: Psoriasis
Keywords: Psoriasis; Immune cell; Cardiovascular; 13N-ammonia; 11C-acetate; Natural History
MeSH Terms: conditions — Psoriasis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Affected Subjects: Subjects diagnosed with moderate- severe psoriasis
  Interventions: Drug: 13N Amonia
- Healthy Controls: Females and males 18 years of age or older

INTERVENTIONS:
Drug: 13N Amonia — Administered during PET/CT scans
  Groups: Affected Subjects

SUMMARY:
Background:

Heart failure (HF) is a public health burden. Studies have shown a link between inflammation, myocardial dysfunction, and HF. Researchers want to use psoriasis as a disease model of chronic inflammation to further study the link between inflammation and myocardial dysfunction.

Objective:

To learn if chronic inflammation affects the heart and if taking a biological medicine for chronic inflammation helps improve how the heart works.

Eligibility:

Adults ages 18 and older who have moderate to severe psoriasis, and healthy adult volunteers.

Design:

Participants will be screened with a medical history. They may take a pregnancy test.

Healthy volunteers will have 1 visit. Those with psoriasis will have a second visit 1 year later.

Participants may give blood samples. They may have a heart function test. They may have a heart imaging test, and may get a contrast agent. If so, it will be injected into a vein.

Participants may have positron emission tomography/computed tomography tests. They will lie on their back on a padded table with their arms straight overhead. They may get radioactive drugs through an intravenous (IV) catheter. They will get stress medicines through the IV. These drugs mimic exercise and increase blood flow through the heart.

Participants may have cardiac magnetic resonance imaging. The scanner is a large tube. Participants will lie on a table that slides in and out of the tube. They will get gadolinium contrast in a vein to improve the pictures. They may get stress medicines. Coils will be used to help make the pictures.

Participation for healthy volunteers will last 1-2 days. Participation for those with psoriasis will last 14 months.

...

DETAILED DESCRIPTION:
Study Description:

Heart failure (HF) remains a significant public health burden despite expanding and improving treatment options. Clinical and pre-clinical studies have demonstrated compelling relationships between inflammation, myocardial dysfunction, HF and adverse clinical outcomes. In this study to be conducted at the NIH Clinical Center, we propose to utilize psoriasis as a disease model to study how chronic inflammation effects myocardial perfusion, measured by myocardial flow reserve (MFR) on positron emission tomography (PET) and cardiac MRI (CMR), and myocardial function and tissue composition measured by multi-modality cardiovascular imaging.

Objectives:

1. To test the hypothesis that chronic inflammation is a driver of perturbances in myocardial perfusion, function, and tissue composition
2. To test the hypothesis that biologic treatment for psoriasis will be associated with longitudinal improvement in myocardial perfusion, function, and tissue composition
3. To characterize immune cell subsets and their association with myocardial perfusion, function, and tissue composition in chronic inflammation
4. To explore how chronic inflammation may alter myocardial energetics and metabolism

Endpoints:

Primary outcomes will be:

Myocardial perfusion, as assessed by myocardial flow reserve (MFR), in subjects with moderate to severe psoriasis compared to matched healthy controls.

Secondary outcomes will be:

Change in MFR in subjects with psoriasis on biologic therapy at 1 year follow-up compared to baseline.

Diastolic function (on echocardiogram), myocardial mechanics (on echocardiogram and CMR), myocardial edema and inflammation, and interstitial fibrosis (on CMR) in subjects with moderate to severe psoriasis compared to matched healthy controls.

Change in diastolic function, myocardial mechanics, myocardial edema and inflammation, and interstitial fibrosis in subjects with psoriasis on biologic therapy at 1 year follow- up

Exploratory outcomes will be:

Immune cell subsets by flow cytometry in subjects with 7 moderate to severe psoriasis compared to matched healthy controls

Rest and stress left ventricular oxygen consumption (MVO2) in subjects with moderate to severe psoriasis compared to matched healthy controls

ELIGIBILITY:
* INCLUSION CRITERIA:

Subjects of both genders will be considered for inclusion in this study. There will be no racial, ethnic, or gender discrimination.

Affected Subjects:

* 18 years of age or older
* Diagnosed with moderate-severe psoriasis clinically confirmed by a licensed physician, or advanced practitioner consisting of typical skin findings and/or associated findings of systemic disease of joints, nails, and hair and may be scheduled to initiate biologic

treatment for psoriasis

Healthy Controls:

Females and males 18 years of age or older

EXCLUSION CRITERIA:

Affected Subjects:

* Pregnant or lactating women
* Subjects with a contraindication to MRI scanning will not receive the CMR assessment.

These contraindications include subjects with the following devices:

i. Central nervous system aneurysm clips

ii. Implanted neural stimulator

iii. Implanted cardiac pacemaker or defibrillator

iv. Cochlear implant

v. Ocular foreign body (e.g. metal shavings)

vi. Implanted Insulin pump

vii. Metal shrapnel or bullet

viii. Estimated glomerular filtration rate (eGFR) < 30 mL/min/1.73m^2 body surface area according to the Modification of Diet in Renal Disease criteria

* History of seizures or taking anti-epileptic medications
* Inability to provide informed consent

Healthy Controls:

* Diagnosis of inflammatory disease (including psoriasis, psoriatic arthritis, rheumatoid arthritis, lupus, inflammatory bowel disease)
* Pregnant women and lactating women
* Subjects with a contraindication to MRI scanning will not receive the CMR assessment.

These contraindications include subjects with the following devices:

ix. Central nervous system aneurysm clips

x. Implanted neural stimulator

xi. Implanted cardiac pacemaker or defibrillator

xii. Cochlear implant

xiii. Ocular foreign body (e.g. metal shavings)

xiv. Implanted Insulin pump

xv. Metal shrapnel or bullet

xvi. Estimated glomerular filtration rate (eGFR) < 30 mL/min/1.73m^2 body surface area according to the Modification of Diet in Renal Disease criteria

* History of seizures or taking anti-epileptic medications
* Inability to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: This is a primary clinical protocol. Affected subjects are defined as patients whose psoriasis is diagnosed clinically by a referring dermatologist or rheumatologist, some of which are planning to start biologic therapy for psoriasis. Healthy controls are also enrolled from the community.
Sampling Method: Non-Probability Sample
Enrollment: 16 (Actual)
Dates: Start 2021-06-07 (Actual); Primary Completion 2022-05-06 (Actual); Study Completion 2022-05-18 (Actual)

PRIMARY OUTCOMES:
Miocardial perfusion in affected vs healthy individuals | 1 day
  Primary outcome will be: Myocardial perfusion, as assessed by myocardial flow reserve (MFR), in subjects with moderate to severe psoriasis compared to matched healthy controls.

SECONDARY OUTCOMES:
Change in MFR in subjects on biologic therapy | 1 year
  Change in MFR in subjects with psoriasis on biologic therapy at 1 year follow-up compared to baseline. 2.Diastolic function (on echocardiogram), myocardial mechanics (on echocardiogram and CMR), myocardial edema and inflammation, and interstitial fibrosis (on CMR) in subjects with moderate to severe psoriasis compared to matched healthy controls. 3.Change in diastolic function, myocardial mechanics, myocardial edema and inflammation, and interstitial fibrosis in subjects with psoriasis on biologic therapy at 1 year follow- up

CONTACTS AND LOCATIONS:
Overall Officials: Michael N Sack, M.D., Principal Investigator — National Heart, Lung, and Blood Institute (NHLBI)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Undecided
.This is a new requirement.

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_000136-H.html

DOCUMENTS (1):
  • Informed Consent Form (2022-06-28): https://cdn.clinicaltrials.gov/large-docs/27/NCT04870827/ICF_000.pdf